CLINICAL TRIAL: NCT01820806
Title: Investigation of the Pharmacokinetics and Metabolism of GLPG0634 in Healthy Male Subjects Following a Single Oral Administration of [14C] GLPG0634
Brief Title: Investigation of the Pharmacokinetics and Metabolism of GLPG0634 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0634-CL-105
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C] GLPG0634 (Experimental): Subjects will be dosed with a single oral 100 mg dose of [14C] GLPG0634 on one occasion
  Interventions: Drug: 100 mg dose of [14C] GLPG0634

INTERVENTIONS:
Drug: 100 mg dose of [14C] GLPG0634 — Subjects will be dosed with a single oral 100 mg dose of [14C] GLPG0634 on one occasion

SUMMARY:
This will be a study in 6 healthy male subjects, each receiving a single oral dose of 100 mg [14C]-radiolabeled GLPG0634.

The study aims to establish the elimination pathways of GLPG0634 and their relative significance and to assess the metabolite profile of GLPG0634 in plasma and in excreta.

Furthermore, the pharmacokinetics (PK) of the main metabolites in plasma relative to GLPG0634 will be evaluated.

This study will also provide safety and tolerability information for GLPG0634.

ELIGIBILITY:
Inclusion Criteria:

* male, between 40 and 65 years of age, inclusive
* within BMI range 18 to 30 kg/m2, inclusive

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The amount of total radioactivity in urine and faeces over time after a single dose of radiolabeled GLPG0634 | Day -1 (pre-dosing) up to Day 10 post dosing
  To evaluate the mass balance recovery of total radioactivity in urine, faeces, and urine and faeces combined to determine the elimination pathways and their relative significance after a single dose of radiolabeled GLPG0634
The amount of GLPG0634 and its main metabolites in urine and faeces over time after a single dose of radiolabeled GLPG0634 | Day -1 (pre-dosing) up to Day 10 post dosing
  To evaluate the recovery of GLPG0634 and its main metabolites in urine and faeces after a single dose of radiolabeled GLPG0634 to determine the elimination pathways and their relative significance (excretion and renal clearance)
Identification of metabolites over time in plasma, urine and faeces after a single dose of radiolabeled GLPG0634 | Day -1 (pre-dosing) up to Day 10 post dosing
  Metabolite profiling and identification in plasma, urine and faeces over time after a single dose of radiolabeled GLPG0634
The amount of radioactivity, GLPG0634 and its main metabolites in blood and plasma over time after a single dose of radiolabeled GLPG0634 | Day 1 (pre-dosing) up to Day 8 post dosing
  To characterize the amount of radioactivity, GLPG0634 and its main metabolites in blood and plasma over time after a single dose of radiolabeled GLPG0634

SECONDARY OUTCOMES:
Number of adverse events | Screening up to Day 10 post dosing
  To evaluate the safety and tolerability of GLPG0634 after a single dose of radiolabeled GLPG0634 in terms of the number of adverse events reported
Changes in vital signs as measured by heart rate, blood pressure and oral temperature | Screening up to Day 10 post dosing
  To evaluate the safety and tolerability of GLPG0634 after a single dose of radiolabeled GLPG0634 in terms of changes in vital signs as measured by heart rate, blood pressure and oral temperature reported
Changes in 12-lead ECG measures | Screening up to Day 10 post dosing
  To evaluate the safety and tolerability of GLPG0634 after a single dose of radiolabeled GLPG0634 in terms of changes in 12-ECG measures reported
Changes in physical exam measures | Screening up to Day 10 post dosing
  To evaluate the safety and tolerability of GLPG0634 after a single dose of radiolabeled GLPG0634 in terms of changes in physical exam measures reported
Changes in blood safety lab parameters | Screening up to Day 10 post dosing
  To evaluate the safety and tolerability of GLPG0634 after a single dose of radiolabeled GLPG0634 in terms of changes in blood safety lab parameters reported
Changes in urine safety lab parameters | Screening up to Day 10 post dosing
  To evaluate the safety and tolerability of GLPG0634 after a single dose of radiolabeled GLPG0634 in terms of changes in urine safety lab parameters reported

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric - Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom